CLINICAL TRIAL: NCT01997840
Title: A Phase 1B/2 Multi-Center, Open Label, Dose-Escalation Study to Determine the Maximum Tolerated Dose, Safety, and Efficacy of ACY-1215 (RICOLINOSTAT) in Combination With Pomalidomide and Low-Dose Dexamethasone in Patients With Relapsed and Refractory Multiple Myeloma
Brief Title: ACY-1215 (Ricolinostat) in Combination With Pomalidomide and Low-dose Dex in Relapsed-and-Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Change in business priorities.
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACE-MM-102
Record Dates: First submitted 2013-11-20; First posted 2013-11-28 (Estimated); Results first posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Neoplasms, Plasma Cell; Neoplasms by Histologic Type; Neoplasms; Blood Protein Disorders; Hematologic Diseases; Dexamethasone; Dexamethasone acetate; Pomalidomide
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell; Neoplasms by Histologic Type; Neoplasms; Blood Protein Disorders; Hematologic Diseases | interventions — ricolinostat; pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ACY-1215 in combination with pomalidomide and dexamethasone (Experimental): ACY-1215 (Ricolinostat) in combination with pomalidomide and dexamethasone
  Interventions: Drug: ACY-1215 (Ricolinostat) in combination with pomalidomide and dexamethasone

INTERVENTIONS:
Drug: ACY-1215 (Ricolinostat) in combination with pomalidomide and dexamethasone — ACY-1215 (Ricolinostat) 160mg QD Days 1-21 with pomalidomide 4mg QD Days 1-21 and dexamethasone 40mg QD Days 1,8,15,22 of a 28-day cycle
  Other Names: Pomalyst; Ricolinostat; Dexamethasone

SUMMARY:
Phase 1b: To evaluate the side effects and determine the best dose of ACY-1215 in combination with Pomalidomide and low-dose dexamethasone in patients with relapsed-and-refractory multiple myeloma.

Phase 2: To determine the overall response rate of ACY-1215 in combination with Pomolidomide and low-dose dexamethasone in patients with relapsed-and-refractory multiple myeloma

ELIGIBILITY:
Inclusion Criteria:

* Must have a documented diagnosis of multiple myeloma and have relapsed-and-refractory disease. Patients must have received at least 2 lines of prior therapies. Patients must have relapsed after having achieved at least stable disease (SD) for at least one cycle of treatment to at least one prior regimen and then developed progressive disease (PD). Patients must also have documented evidence of PD during or within 60 days (measured from the end of the last cycle) of completing treatment with the last anti-myeloma drug regimen used just prior to study entry (refractory disease)
* Must have undergone prior treatment with at least 2 cycles of lenalidomide and at least 2 cycles of a proteasome inhibitor (either in separate regimens or within the same regimen)
* Must not be a candidate for autologous stem cell transplant (ASCT), has declined the option of ASCT, or has relapsed after prior ASCT
* Must have measurable levels of myeloma paraprotein in serum (≥ 0.5 g/dL) or urine (≥ 0.2 g/24 hours)
* Must have Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2
* Females of child bearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10 - 14 days prior to, and again within 24 hours of starting pomalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking pomalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a vasectomy. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure. Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods,and Education and Counseling Guidance must be followed per protocol
* Must be able to take acetylsalicylic acid (ASA) (81 or 325 mg) daily as prophylactic anticoagulation. Patients intolerant to ASA may use low molecular weight heparin. Lovenox is recommended. Coumadin will be allowed provided the patient is fully anticoagulated, with an international normalized ratio (INR) of 2 to 3

Exclusion Criteria:

* Pregnant or lactating females
* Prior therapy with HDAC inhibitor
* Any of the following laboratory abnormalities:

  * ANC < 1,000/µL
  * Platelet count < 75,000/ µL for patients in whom < 50% of bone marrow nucleated cells are plasma cells; and < 50,000/ µL for patients in whom ≥ 50% of bone marrow nucleated cells are plasma cells
  * Hemoglobin < 8g/dL (<4.9 mmol/L; prior red blood cell [RBC] transfusion is permitted)
  * Creatine clearance < 45mL/min according to Cockcroft-Gault formula. If creatine clearance calculated from the 24-hour urine sample is ≥ 45 mL/min, patient will qualify for the study
  * Serum glutamic oxaloacetic transaminase (SGOT)/aspartate aminotransferase (AST), or serum glutamic pyruvic transaminase (SGPT)/ alanine aminotransferase (ALT) > 3.0 × ULN
  * Serum total bilirubin > 2.0 mg/dL
* Prior history of malignancies, other than MM, unless the patient has been free of the disease for ≥ 3 years. Exceptions include the following:

  * Basal or squamous cell carcinoma of the skin
  * Carcinoma in situ of the cervix or breast
  * Incidental histologic finding of prostate cancer (TNM stage of T1a or T1b)
* Corrected QT interval using Fridericia's formula (QTcF) value > 480 msec at screening; family or personal history of long QTc syndrome or ventricular arrhythmias including ventricular bigeminy; previous history of drug-induced QTc prolongation or the need for treatment with medications known or suspected of producing prolonged QTc intervals on electrocardiogram (ECG)
* Positive human immunodeficiency virus (HIV), hepatitis B virus (HBV) and/or hepatitis C virus (HCV) infection
* Hypersensitivity to thalidomide, lenalidomide, or dexamethasone (such as Steven Johnson Syndrome). Hypersensitivity, such as rash, that can be medically managed is allowable
* Peripheral neuropathy ≥ Grade 2 despite supportive therapy
* Radiotherapy or systemic therapy (standard or an investigational or biologic anticancer agent) within 14 days of initiation of study drug treatment
* Current enrollment in another clinical trial involving treatment and/or is receiving an investigational agent for any reason
* Inability or unwillingness to comply with birth control requirements or regional REMS/RevAid programs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- United States (2):
  - Local Institution - 201, Boston, Massachusetts
  - Cleveland Clinic, Cleveland, Ohio

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of Phase 1b (dose finding segment) part and Phase 2(dose expansion segment) part.
Groups:
- Phase 1b - ACY-1215 Dose Level 1; Phase 2 - ACY-1215 Dose Level 1: Participants received 160 mg ACY-1215 and 4 mg pomalidomide daily on Days 1-21 of each 28-day cycle. Participants also received 40 mg (<=75 years) or 20 mg (>75 years) dexamethasone on Days 1, 8, 15, and 22 of each 28-day treatment cycle.
- Phase 1b - ACY-1215 Dose Level 3; Phase 2 - ACY-1215 Dose Level 3: Participants received 160 mg ACY-1215 twice daily in combination with 4 mg pomalidomide once daily on Days 1-21 of each 28-day cycle. Participants also received 40 mg (<=75 years) or 20 mg (>75 years) dexamethasone on Days 1, 8, 15, and 22 of each 28-day treatment cycle.
Period: Overall Study
Arm/Group | Phase 1b - ACY-1215 Dose Level 1 | Phase 1b - ACY-1215 Dose Level 3 | Phase 2 - ACY-1215 Dose Level 1 | Phase 2 - ACY-1215 Dose Level 3
Started (Started treatment) | 3 | 4 | 85 | 11
Efficacy Evaluable Population | 3 | 4 | 77 | 7
Safety Population | 3 | 4 | 85 | 11
Completed | 0 | 0 | 0 | 0
Not Completed | 3 | 4 | 85 | 11
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Withdrawal by participant | 0 | 0 | 8 | 1
Not completed — Physician Decision | 0 | 0 | 3 | 0
Not completed — Progressive disease | 3 | 4 | 57 | 8
Not completed — Other reasons | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 15 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1b - ACY-1215 Dose Level 1 | Phase 1b - ACY-1215 Dose Level 3 | Phase 2 - ACY-1215 Dose Level 1 | Phase 2 - ACY-1215 Dose Level 3 | Total
Number analyzed (Participants) | 3 | 4 | 85 | 11 | 103
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 42 | 4 | 50
  >=65 years | 1 | 2 | 43 | 7 | 53
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 40 | 4 | 47
  Male | 1 | 3 | 45 | 7 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 3 | 4 | 81 | 11 | 99
  Unknown or Not Reported | 0 | 0 | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 7 | 1 | 8
  White | 3 | 4 | 72 | 10 | 89
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of ACY-1215- Phase 1b
Description: The maximum tolerated dose (MTD) was defined as the highest dose level at which no more than 1 of 6 patients experienced a dose-limiting toxicity (DLT) within the first 28-day cycle. If no more than 1 of these 6 patients experienced a DLT within the first 28-day cycle, then the last dose level enrolled to meet these criteria was identified as the recommended dose for the Phase 2 segment of the study.
Time Frame: From first dose until the end of Phase 1b (up to a maximum of approximately 50 weeks).
Population: All treated participants in Phase 1b. Prespecified to be reported as combined for Phase 1b only.
Measure: Number; unit: mg/day
Groups:
- Phase 1b - ACY-1215: Participants received either 160 mg ACY-1215 once per day (Dose Level 1) or 160 mg ACY-1215 twice per day (Dose Level 3) and 4 mg pomalidomide daily on Days 1-21 of each 28-day cycle. Participants also received 40 mg (<=75 years) or 20 mg (>75 years) dexamethasone on Days 1, 8, 15, and 22 of each 28-day treatment cycle.
Arm/Group | Phase 1b - ACY-1215
Number analyzed (Participants) | 7
mg/day | 320

2. Primary Outcome: Overall Response Rate (ORR) Per Investigator - Phase 2
Description: Overall response rate (ORR) is defined as the percentage of participants with a best response of stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR).
  sCR:
  * No detectable myeloma cells in the bone marrow.
  * Normal free light chain ratio.
  * Absence of clonal cells in the bone marrow.
  CR:
  * Negative immunofixation on the serum and urine.
  * Disappearance of any soft tissue plasmacytomas.
  * Less than 5% plasma cells in the bone marrow.
  VGPR:
  * Serum and urine M-protein detectable by immunofixation but not on electrophoresis, or
  * At least a 90% reduction in serum M-protein plus urine M-protein level less than 100 mg per 24 hours.
  PR:
  * At least a 50% reduction in serum M-protein.
  * Reduction in 24-hour urinary M-protein by at least 90% or to less than 200 mg per 24 hours.
  * For patients with non-secretory myeloma, a reduction of at least 50% in the size of soft tissue plasmacytomas is required.
Time Frame: From first dose until disease progression, study drug toxicity, end of study, or death due to any cause (up to approximately 120 months).
Population: All treated participants in Phase 2 Efficacy evaluable population. Prespecified to be reported for Phase 2 only.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Phase 2 - ACY-1215 Dose Level 1 | Phase 2 - ACY-1215 Dose Level 3
Number analyzed (Participants) | 77 | 7
Percent of Participants | 39.0 [28.0 to 50.8] | 71.4 [29.0 to 96.3]

3. Secondary Outcome: Time to Response (TTR)
Description: Time to response (TTR) was defined as the time from first dose of study treatment to the first documentation of response (either partial response (PR) or complete response (CR)).
  CR:
  * Negative immunofixation on the serum and urine.
  * Disappearance of any soft tissue plasmacytomas.
  * Less than 5% plasma cells in the bone marrow.
  PR:
  * At least a 50% reduction in serum M-protein.
  * Reduction in 24-hour urinary M-protein by at least 90% or to less than 200 mg per 24 hours.
  * For patients with non-secretory myeloma, a reduction of at least 50% in the size of soft tissue plasmacytomas is required.
Time Frame: as for outcome 2
Population: All treated participants in the Efficacy Evaluable population with a best response of PR or CR.
Measure: Mean (Full Range); unit: Weeks
Arm/Group | Phase 1b - ACY-1215 Dose Level 1 | Phase 1b - ACY-1215 Dose Level 3 | Phase 2 - ACY-1215 Dose Level 1 | Phase 2 - ACY-1215 Dose Level 3
Number analyzed (Participants) | 2 | 0 | 30 | 5
Weeks | 8.50 [4.1 to 12.9] |  | 10.83 [4.1 to 40.1] | 12.96 [7.9 to 31.9]

4. Secondary Outcome: Duration of Response (DoR)
Description: Duration of Response (DOR) was defined as the time from first partial response (PR) or complete response (CR) to the first documentation of progressive disease (PD) or death.
  PR:
  * >= 50% reduction in serum M-protein.
  * Reduction in 24-hour urinary M-protein by >= 90% or to less than 200 mg per 24 hours.
  * For non-secretory myeloma, a reduction of >= 50% in size of soft tissue plasmacytomas.
  CR:
  * Negative immunofixation on the serum and urine.
  * Disappearance of any soft tissue plasmacytomas.
  * < 5% plasma cells in the bone marrow.
  PD:
  * Increase of 25% or more from nadir in serum M-protein, absolute increase of >= 0.5 g/dL.
  * Increase of 25% or more from nadir in 24-hour urinary M-protein, absolute increase of >=200 mg/24 hours.
  * Increase of 25% or more in the percentage of bone marrow plasma cells, absolute increase of >=10%.
  Calculated using Kaplan-Meier estimates.
Time Frame: as for outcome 2
Population: All treated participants in the Efficacy Evaluable population with a best response of PR or CR.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Phase 1b - ACY-1215 Dose Level 1 | Phase 1b - ACY-1215 Dose Level 3 | Phase 2 - ACY-1215 Dose Level 1 | Phase 2 - ACY-1215 Dose Level 3
Number analyzed (Participants) | 2 | 0 | 30 | 5
Weeks | 20.10 [4.10 to 36.10] |  | 30.30 [13.10 to 43.10] | 62.75 [54.75 to 121.6]

5. Secondary Outcome: Time to Progression (TTP)
Description: Time to progression (TTP) was defined as the time from the date of first dose to the date of first documentation of progressive disease (PD).
  PD:
  * Increase of 25% or more from nadir in serum M-protein, absolute increase of >= 0.5 g/dL.
  * Increase of 25% or more from nadir in 24-hour urinary M-protein, absolute increase of >=200 mg/24 hours.
  * Increase of 25% or more in the percentage of bone marrow plasma cells, absolute increase of >=10%.
  * New bone lesions or soft tissue plasmacytomas or increase size of existing bone lesions or soft tissue plasmacytomas.
  * Hypercalcemia attributed to myeloma.
Time Frame: as for outcome 2
Population: All treated participants in the Efficacy Evaluable population who had PD.
Measure: Mean (Full Range); unit: Weeks
Arm/Group | Phase 1b - ACY-1215 Dose Level 1 | Phase 1b - ACY-1215 Dose Level 3 | Phase 2 - ACY-1215 Dose Level 1 | Phase 2 - ACY-1215 Dose Level 3
Number analyzed (Participants) | 3 | 4 | 77 | 7
Weeks | 22.43 [8.1 to 48.9] | 6.20 [4.1 to 8.1] | 29.82 [3.9 to 169.1] | 83.22 [7.7 to 183.1]

6. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) was defined as the time from first dose of study treatment to the first documentation of progressive disease (PD) or death from any cause during study
  PD:
  * Increase of 25% or more from nadir in serum M-protein, absolute increase of >= 0.5 g/dL.
  * Increase of 25% or more from nadir in 24-hour urinary M-protein, absolute increase of >=200 mg/24 hours.
  * Increase of 25% or more in the percentage of bone marrow plasma cells, absolute increase of >=10%.
  * New bone lesions or soft tissue plasmacytomas or increase size of existing bone lesions or soft tissue plasmacytomas.
  * Hypercalcemia attributed to myeloma. Calculated using Kaplan-Meier estimates.
Time Frame: as for outcome 2
Population: All treated participants in the Efficacy Evaluable population.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Phase 1b - ACY-1215 Dose Level 1 | Phase 1b - ACY-1215 Dose Level 3 | Phase 2 - ACY-1215 Dose Level 1 | Phase 2 - ACY-1215 Dose Level 3
Number analyzed (Participants) | 3 | 4 | 77 | 7
Weeks | 10.30 [8.10 to 48.90] | 6.30 [4.35 to 8.05] | 20.00 [9.10 to 41.60] | 62.70 [19.90 to 99.90]

7. Secondary Outcome: Overall Response Rate (ORR) Per Central Adjudication Committee
Description: Overall response rate (ORR) per Central Adjudication Committee is the percentage of participants with a best response of stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR).
  sCR:
  * No detectable myeloma cells in the bone marrow.
  * Normal free light chain ratio.
  * Absence of clonal cells in the bone marrow.
  CR:
  * Negative immunofixation on the serum and urine.
  * Disappearance of any soft tissue plasmacytomas.
  * Less than 5% plasma cells in the bone marrow.
  VGPR:
  * Serum and urine M-protein detectable by immunofixation but not on electrophoresis, or
  * At least a 90% reduction in serum M-protein plus urine M-protein level less than 100 mg per 24 hours.
  PR:
  * At least a 50% reduction in serum M-protein.
  * Reduction in 24-hour urinary M-protein by at least 90% or to less than 200 mg per 24 hours.
  * For patients with non-secretory myeloma, a reduction of at least 50% in the size of soft tissue plasmacytomas is required
Time Frame: as for outcome 2
Population: All treated participants in the Efficacy Evaluable population. Data not collected.
Arm/Group | Phase 1b - ACY-1215 Dose Level 1 | Phase 1b - ACY-1215 Dose Level 3 | Phase 2 - ACY-1215 Dose Level 1 | Phase 2 - ACY-1215 Dose Level 3
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An adverse event (AE) is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a participant during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the participant's health, including laboratory test values, regardless of etiology. Any worsening (i.e., any clinically significant adverse change in the frequency or intensity of a preexisting condition) should be considered an AE. Graded according to NCI CTCAE (Version 4.03) guidelines where grade 1 = mild, grade 2 = moderate, grade 3 = severe, grade 4 = life threatening, grade 5 = death.
Time Frame: From first dose until 30 days after last dose of study drug (assessed for an average of approximately 55 weeks to a maximum of approximately 456 weeks)
Population: All treated participants in the Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b - ACY-1215 Dose Level 1 | Phase 1b - ACY-1215 Dose Level 3 | Phase 2 - ACY-1215 Dose Level 1 | Phase 2 - ACY-1215 Dose Level 3
Number analyzed (Participants) | 3 | 4 | 85 | 11
Participants | 3 | 4 | 82 | 11

9. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: A serious adverse event (SAE) is defined as any adverse event (AE) occurring at any dose that:
  * Results in death;
  * Is life-threatening (ie, in the opinion of the Investigator, the participant is at immediate risk of death from the AE);
  * Requires inpatient hospitalization or prolongation of existing hospitalization (hospitalization is defined as an inpatient admission, regardless of length of stay).
  * Results in persistent or significant disability/incapacity (a substantial disruption of the participant's ability to conduct normal life functions);
  * Is a congenital anomaly/birth defect;
  * Constitutes an important medical event. Graded according to NCI CTCAE (Version 4) guidelines where grade 1 = mild, grade 2 = moderate, grade 3 = severe, grade 4 = life threatening, grade 5 = death.
Time Frame: as for outcome 8
Population: All treated participants in the Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b - ACY-1215 Dose Level 1 | Phase 1b - ACY-1215 Dose Level 3 | Phase 2 - ACY-1215 Dose Level 1 | Phase 2 - ACY-1215 Dose Level 3
Number analyzed (Participants) | 3 | 4 | 85 | 11
Participants | 0 | 2 | 37 | 7

10. Secondary Outcome: Number of Participants With Adverse Events (AEs) Leading to Discontinuation
Description: as for outcome 8
Time Frame: as for outcome 8
Population: All treated participants in the Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b - ACY-1215 Dose Level 1 | Phase 1b - ACY-1215 Dose Level 3 | Phase 2 - ACY-1215 Dose Level 1 | Phase 2 - ACY-1215 Dose Level 3
Number analyzed (Participants) | 3 | 4 | 85 | 11
Participants
  ACY-1215 | 0 | 0 | 13 | 1
  Pomalidomide | 0 | 0 | 13 | 1
  Dexamethasone | 0 | 0 | 16 | 1

11. Secondary Outcome: Number of Participants With Adverse Events (AEs) Related to Study Drug
Description: as for outcome 8
Time Frame: as for outcome 8
Population: All treated participants in the Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b - ACY-1215 Dose Level 1 | Phase 1b - ACY-1215 Dose Level 3 | Phase 2 - ACY-1215 Dose Level 1 | Phase 2 - ACY-1215 Dose Level 3
Number analyzed (Participants) | 3 | 4 | 85 | 11
Participants
  ACY-1215 | 1 | 4 | 63 | 9
  Pomalidomide | 3 | 4 | 62 | 11
  Dexamethasone | 2 | 3 | 57 | 9

12. Secondary Outcome: Plasma Levels of ACY-1215 and Pomalidomide - Phase 1b
Time Frame: Cycle 1 day 1, Cycle 1 Day 2, Cycle 1 Day 8
Population: All treated participants with available PK results. Prespecified to be reported for Phase 1b only. Data not collected.
Arm/Group | Phase 1b - ACY-1215 Dose Level 1 | Phase 1b - ACY-1215 Dose Level 3
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADA) - Phase 1b
Time Frame: Cycle 1 day 1, Cycle 1 Day 2, Cycle 1 Day 8
Population: All treated participants with available ADA results. Prespecified to be reported for Phase 1b only. Data not collected.
Arm/Group | Phase 1b - ACY-1215 Dose Level 1 | Phase 1b - ACY-1215 Dose Level 3
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Participants were assessed for All-Cause Mortality from first dose until study completion (assessed up to approximately 120 months). SAEs and Other AEs were assessed from first dose until 30 days after last dose of study drug (assessed for an average of approximately 55 weeks to a maximum of approximately 456 weeks).
Description: All-Cause Mortality, Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication.
Arm/Group | Phase 1b - ACY-1215 Dose Level 1 | Phase 1b - ACY-1215 Dose Level 3 | Phase 2 - ACY-1215 Dose Level 1 | Phase 2 - ACY-1215 Dose Level 3
All-Cause Mortality (participants affected / at risk) | 2/3 | 1/4 | 39/85 | 3/11
Serious Adverse Events (participants affected / at risk) | 0/3 | 2/4 | 37/85 | 7/11
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 82/85 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b - ACY-1215 Dose Level 1 (N=3) | Phase 1b - ACY-1215 Dose Level 3 (N=4) | Phase 2 - ACY-1215 Dose Level 1 (N=85) | Phase 2 - ACY-1215 Dose Level 3 (N=11)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 1 | 0
Sudden death (General disorders) | 0 | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 2 | 0
Corona virus infection (Infections and infestations) | 0 | 0 | 1 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Haemophilus infection (Infections and infestations) | 0 | 0 | 1 | 0
Implant site infection (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Meningitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 6 | 2
Pneumonia parainfluenzae viral (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia viral (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 0
Sepsis (Infections and infestations) | 0 | 0 | 3 | 0
Septic shock (Infections and infestations) | 0 | 0 | 2 | 0
Streptococcal bacteraemia (Infections and infestations) | 0 | 0 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 3 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0
Embolic stroke (Nervous system disorders) | 0 | 0 | 1 | 0
Radiculopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 2 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b - ACY-1215 Dose Level 1 (N=3) | Phase 1b - ACY-1215 Dose Level 3 (N=4) | Phase 2 - ACY-1215 Dose Level 1 (N=85) | Phase 2 - ACY-1215 Dose Level 3 (N=11)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 31 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 29 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 17 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 2
Sinus tachycardia (Cardiac disorders) | 1 | 1 | 1 | 0
Tricuspid valve disease (Cardiac disorders) | 0 | 0 | 0 | 1
Deafness (Ear and labyrinth disorders) | 0 | 0 | 1 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 1
Cushingoid (Endocrine disorders) | 0 | 0 | 2 | 1
Cataract (Eye disorders) | 0 | 0 | 0 | 2
Dacryostenosis acquired (Eye disorders) | 0 | 0 | 0 | 1
Diplopia (Eye disorders) | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 1
Ectropion (Eye disorders) | 0 | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 0 | 1 | 1
Vision blurred (Eye disorders) | 0 | 1 | 3 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 7 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 7 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 6 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 3 | 14 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 4 | 32 | 6
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 4 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 3 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 3 | 2
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 19 | 3
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Sensitivity of teeth (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 9 | 1
Asthenia (General disorders) | 0 | 1 | 7 | 0
Chest discomfort (General disorders) | 0 | 0 | 1 | 1
Chest pain (General disorders) | 0 | 1 | 4 | 0
Chills (General disorders) | 0 | 1 | 4 | 1
Fatigue (General disorders) | 2 | 2 | 49 | 8
Feeling jittery (General disorders) | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 5 | 0
Instillation site pain (General disorders) | 0 | 1 | 4 | 2
Local swelling (General disorders) | 0 | 0 | 4 | 2
Oedema (General disorders) | 0 | 0 | 5 | 0
Oedema peripheral (General disorders) | 0 | 0 | 13 | 2
Pyrexia (General disorders) | 0 | 1 | 18 | 1
Vessel puncture site bruise (General disorders) | 0 | 1 | 0 | 0
Hypogammaglobulinaemia (Immune system disorders) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 3 | 2
Gastroenteritis (Infections and infestations) | 0 | 0 | 3 | 1
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 1
Herpes virus infection (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 3 | 2
Localised infection (Infections and infestations) | 0 | 0 | 3 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 8 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 21 | 3
Urinary tract infection (Infections and infestations) | 0 | 0 | 6 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 2
Periorbital contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Scar (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 7 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 6 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 4 | 0
Blood cholesterol increased (Investigations) | 1 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 7 | 2
Blood glucose increased (Investigations) | 0 | 0 | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0
Haematocrit decreased (Investigations) | 0 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 3 | 0 | 0 | 3
Lymphocyte count decreased (Investigations) | 0 | 0 | 2 | 1
Neutrophil count decreased (Investigations) | 2 | 1 | 12 | 3
Platelet count decreased (Investigations) | 1 | 0 | 6 | 4
Weight decreased (Investigations) | 0 | 0 | 3 | 2
White blood cell count decreased (Investigations) | 2 | 0 | 4 | 4
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 9 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 2 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 4 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 7 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 4 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 5 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 11 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 3 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1 | 7 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 7 | 2
Polydipsia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 13 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 13 | 3
Bone disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 11 | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 17 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 9 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 9 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 11 | 2
Dizziness postural (Nervous system disorders) | 0 | 0 | 2 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 11 | 1
Headache (Nervous system disorders) | 1 | 0 | 7 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 3 | 1
Memory impairment (Nervous system disorders) | 0 | 0 | 4 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 1 | 4 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 2 | 1
Tremor (Nervous system disorders) | 0 | 0 | 10 | 0
VIth nerve paralysis (Nervous system disorders) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 2 | 2
Confusional state (Psychiatric disorders) | 1 | 0 | 3 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 6 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 16 | 3
Mood altered (Psychiatric disorders) | 1 | 0 | 4 | 2
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 15 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 8 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 9 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 8 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 4 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 8 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 5 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 3
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 5 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 10 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Aortic arteriosclerosis (Vascular disorders) | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 0 | 5 | 0
Hypertension (Vascular disorders) | 2 | 0 | 2 | 4
Hypotension (Vascular disorders) | 0 | 1 | 3 | 2
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1
Peripheral coldness (Vascular disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-12): https://cdn.clinicaltrials.gov/large-docs/40/NCT01997840/Prot_SAP_000.pdf